CLINICAL TRIAL: NCT05021978
Title: A Phase 2 Clinical Trial Evaluating the Efficacy, Safety, Tolerability, and Pharmacokinetics of PRAX-944 in Adults With Essential Tremor
Brief Title: A Clinical Trial of PRAX-944 in Participants With Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAX-944-221
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-01

CONDITIONS: Essential Tremor
Keywords: Movement Disorder; Benign Essential Tremor; Familial Tremor; Hereditary Essential Tremor; Movement Disorder Agents; Calcium Channels, T-type
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Intervention Model Description: Part A: Single group Part B: Parallel group, randomized withdrawal
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A: Open label Part B: Open label titration followed by quadruple-blind, randomized withdrawal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Open-label 20 and 40 mg PRAX-944 (Experimental): Once daily, oral dosing with 7 days of 20 mg and 7 days of 40 mg
  Interventions: Drug: Part A: 20 and 40 mg PRAX-944
- Part B: Open-label titration PRAX-944 (120 mg) followed by blinded PRAX-944 (Experimental): Once daily, oral dosing with titration to 120 mg: 3 days of 20 mg, 4 days of 40 mg, 7 days of 60 mg, 7 days of 80 mg, 7 days of 100 mg, 28 days of 120 mg
  Interventions: Drug: Part B: 120 mg PRAX-944
- Part B: Open-label titration PRAX-944 (120 mg) followed by blinded placebo (Active Comparator): Once daily, oral dosing with titration to 120 mg: 3 days of 20 mg, 4 days of 40 mg, 7 days of 60 mg, 7 days of 80 mg, 7 days of 100 mg, 14 days of 120 mg, 14 days placebo
  Interventions: Drug: Part B: 120 mg PRAX-944 and Placebo

INTERVENTIONS:
Drug: Part A: 20 and 40 mg PRAX-944 — Once daily oral treatment
  Arms: Part A: Open-label 20 and 40 mg PRAX-944
Drug: Part B: 120 mg PRAX-944 — Once daily oral treatment with titration
  Arms: Part B: Open-label titration PRAX-944 (120 mg) followed by blinded PRAX-944
Drug: Part B: 120 mg PRAX-944 and Placebo — Once daily oral treatment with titration followed by placebo
  Arms: Part B: Open-label titration PRAX-944 (120 mg) followed by blinded placebo

SUMMARY:
This is a 2-part clinical trial to evaluate the efficacy, safety, and tolerability of 40 and 120 mg oral PRAX-944 compared to placebo in the treatment of adults with essential tremor. Part A is designed to study the dose titration from 20 to 40 mg every morning (QAM) (ie, 2 weeks with 7 days at each dose level). Part B is designed to study the dose titration from 20 to up to 120 mg QAM with at least 14 days of dosing at the highest tolerated dose for each participant. Blood levels of PRAX-944 will also be measured throughout the trial and pharmacokinetics will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ET consistent with Movement Disorders Society Criteria, a duration of ET of at least 3 years and with onset before the age of 65
2. TETRAS upper limb score (ie, sum of bilateral upper limb items 4a, 4b, and 4c) of ≥10 as rated by the Investigator at Screening and Baseline OR A score of ≥2 on 2 or more of the following TETRAS activities of daily living (ADL) subscale items: (2) Feeding with a spoon, (3) Drinking from a glass, (5) Dressing, (6) Pouring, (9) Writing OR A score of ≥2 on 1 of the following TETRAS ADL subscale items: (2) Feeding with a spoon, (3) Drinking from a glass, (5) Dressing, (6) Pouring, or (9) Writing AND a score of ≥2 on both of the following TETRAS ADL subscale items: (10) Working and (12) Social Impact
3. If currently receiving any medication for ET, is on a stable dose of any of these medications for ET for 28 days prior to Screening and is willing to maintain stable doses throughout the trial. If receiving primidone for ET, is willing and able to discontinue 14 days prior to Day 1.
4. Body mass index (BMI) between 18 and 40 kg/m2 (inclusive).

Exclusion Criteria:

1. Sporadically using a benzodiazepine, sleep medication, or anxiolytic that would confound the assessment of tremor.
2. Trauma to the nervous system within 3 months preceding the onset of tremor.
3. History of other medical, neurological or psychiatric condition that may explain or cause tremor, including but not limited to Parkinson's disease, dystonia, cerebellar disease, family history of Fragile X syndrome, traumatic brain injury, alcohol abuse or withdrawal, benzodiazepine abuse or withdrawal, multiple sclerosis, polyneuropathy, and endocrine states such as hyperthyroidism.
4. Prior magnetic resonance-guided focused ultrasound or surgical intervention for ET such as deep brain stimulation or thalamotomy.
5. Botulinum toxin injection for ET in the 6 months prior to Screening.
6. Unwilling or unable to refrain from alcohol 24 hours before and during clinical trial visits.
7. History of substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Development, Study Director — Praxis Precision Medicines
Locations (9):
- United States (2):
  - Praxis Research Site, Port Charlotte, Florida
  - Praxis Research Site, Spokane, Washington
- Australia (5):
  - Praxis Research Site, New Lambton Heights, New South Whales
  - Praxis Research Site, Southport, Queensland
  - Praxis Research Site, Fitzroy, Victoria
  - Praxis Research Site, Melbourne, Victoria
  - Praxis Research Site, Parkville, Victoria
- New Zealand (2):
  - Praxis Research Site, Grafton, Auckland
  - Praxis Research Site, Christchurch

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: PRAX-944 20mg to 40mg Open-Label Titration (OLT): Participants in open-label titration phase were administered once daily oral dose of PRAX-944 titrated from 20 mg (7 days) to 40 mg (7 days).
- Part B: PRAX-944 20mg to 120mg OLT: Participants in open-label titration phase were administered once daily oral dose of PRAX-944 titrated from 20 mg to up to 120 mg for 6-weeks.
- Part B: PRAX-944 120mg Randomized Withdrawal Phase (RWD): Participants in double-blind, randomized withdrawal phase were administered PRAX-944 120mg for 14 days.
- Part B: Placebo RWD: Participants in double-blind, randomized withdrawal phase were administered Placebo for 14 days.
Period: PART A OLT Phase (Day 1 to Day 21)
Arm/Group | Part A: PRAX-944 20mg to 40mg Open-Label Titration (OLT) | Part B: PRAX-944 20mg to 120mg OLT | Part B: PRAX-944 120mg Randomized Withdrawal Phase (RWD) | Part B: Placebo RWD
Started | 7 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: PART B OLT Phase (Day 1 to Day 42)
Arm/Group | Part A: PRAX-944 20mg to 40mg Open-Label Titration (OLT) | Part B: PRAX-944 20mg to 120mg OLT | Part B: PRAX-944 120mg Randomized Withdrawal Phase (RWD) | Part B: Placebo RWD
Started | 0 | 17 | 0 | 0
Completed | 0 | 11 | 0 | 0
Not Completed | 0 | 6 | 0 | 0
Not completed — Adverse Event | 0 | 6 | 0 | 0
Period: PART B RWD Phase (Day 43 to Day 70)
Arm/Group | Part A: PRAX-944 20mg to 40mg Open-Label Titration (OLT) | Part B: PRAX-944 20mg to 120mg OLT | Part B: PRAX-944 120mg Randomized Withdrawal Phase (RWD) | Part B: Placebo RWD
Started | 0 | 0 | 6 | 5
Completed | 0 | 0 | 6 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: PRAX-944 20mg to 40mg OLT: Participants in open-label titration phase were administered once daily oral dose of PRAX-944 titrated from 20 mg (7 days) to 40 mg (7 days).
- Total: Total of all reporting groups
Arm/Group | Part A: PRAX-944 20mg to 40mg OLT | Part B: PRAX-944 20mg to 120mg OLT | Total
Number analyzed (Participants) | 7 | 17 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (6.60) | 59.3 (13.81) | 61.8 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 14 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 17 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 16 | 22
  More than one race | 0 | 0 | 0
  Aborigines | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Upper Limb Score
Description: The TETRAS upper limb score is calculated as the sum of the 6 separate upper-limb maneuvers assessed by the clinician: forward-outstretched postural tremor [right], forward outstretched postural tremor [left], lateral wing-beating postural tremor [right], lateral wing-beating postural tremor [left], kinetic tremor [right], kinetic tremor [left], each on a 0 (no tremor) to 4 (maximum tremor) severity scale in 0.5-point increments. TETRAS Part 4 score for both upper limbs ranged from 0 to 24, higher scores indicated more severe tremor. A negative change from baseline indicated less tremor. Baseline is defined as the last non-missing value collected prior to receiving first dose of study drug. Change from baseline will be defined as assessment value minus baseline value.
Time Frame: Baseline (Day 0), Days 7 and 14
Population: Full Analysis Set (FAS): all participants who took at least 1 dose of study drug and had a valid baseline TETRAS assessment and at least 1 valid post-baseline TETRAS assessment. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part A: PRAX-944 20mg to 40mg OLT
Number analyzed (Participants) | 6
Scores on a scale
  Change from baseline to Day 7 | -1.427 [-4.4375 to 1.5845]
  Change from baseline to Day 14 | -2.912 [-4.2779 to -1.5466]
Statistical Analysis 1: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Sample size is a convenience sample determined according to feasibility to provide sufficient and safety data to inform the development of future controlled studies with PRAX-944. In the open-label phase of the trial (Part A ), at least 10 participants would provide an 80% probability of observing at least 1 AE with an underlying incidence of 15% or greater and provide approximately 80% power to detect an effect size of 1.0 on the primary endpoint change from baseline in TETRAS Upper Limb score; Test type: Other; p = 0.1048, Mixed Models Analysis — Change from baseline to Day 7 in TETRAS Upper Limb Score; Includes timepoint as fixed effect and baseline TETRAS score as a covariate. Within subject variability modeled using unstructured covariance pattern
Statistical Analysis 2: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.0028, Mixed Models Analysis — Change from baseline to Day 14 in TETRAS UL score

2. Primary Outcome: Part B: Number of Participants With Adverse Events (AE), Related AE, and AE Leading to Treatment Discontinuation
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Incidence and Severity of Adverse Events have been reported.
Time Frame: Up to Day 70
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Part B: PRAX-944 120mg RWD: Participants in double-blind, randomized withdrawal phase were administered PRAX-944 120mg for 14 days.
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT | Part B: PRAX-944 120mg RWD | Part B: Placebo RWD
Number analyzed (Participants) | 17 | 6 | 5
participants
  Any AE | 15 | 1 | 1
  Related AE | 12 | 0 | 1
  AE Leading to Treatment Discontinuation | 6 | 0 | 0
  Mild AE | 13 | 1 | 1
  Moderate AE | 7 | 1 | 0
  Severe AE | 0 | 0 | 1

3. Primary Outcome: Part B: Number of Participants With Clinically Significant Abnormalities in Vital Signs, Laboratory Values and Electrocardiogram Parameters
Description: Vital signs parameters included body temperature, pulse rate, respiratory rate, blood pressure (systolic and diastolic), clinical laboratory measures (chemistry, hematology, urinalysis, and coagulation), electrocardiogram parameters (heart rate, PR, QRS, QT, and corrected QT intervals). Any change in vital sign abnormalities that was clinically significant in the medical and scientific judgment of the investigator and not related to an underlying disease was reported as an unsolicited adverse event (AE). Any clinically significant abnormality associated with underlying disease does not require reporting as an (S)AE unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Day 70
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT | Part B: PRAX-944 120mg RWD | Part B: Placebo RWD
Number analyzed (Participants) | 17 | 6 | 5
participants | 0 | 0 | 0

4. Primary Outcome: Part B: Number of Participants With Suicidal Ideation or Behavior Assessed Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is described as a scale developed at Columbia University that has 2-6 questions each in categories of Suicidal Ideation, Intensity of Ideation, Suicidal Behavior, and Actual Attempts. Four constructs were measured. Severity of Suicidal ideation is rated on a 5-point ordinal scale. Intensity of ideation is comprised of 5 items (frequency, duration, controllability, deterrents, and reason for ideation), each rated on a 5-point ordinal scale. Suicidal behavior is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and non-suicidal self-injurious behavior. Lethality, assesses actual attempts; actual lethality is rated on a 6-point ordinal scale, and if actual lethality is 0, potential lethality of attempts is rated on a 3-point ordinal scale.The higher the C-SSRS score, the higher the suicide risk (ie. worse outcome).
Time Frame: Up to Day 70
Population: FAS population
Measure: Number; unit: Participants
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT | Part B: PRAX-944 120mg RWD | Part B: Placebo RWD
Number analyzed (Participants) | 17 | 6 | 5
Participants | 0 | 0 | 0

5. Secondary Outcome: Part A: Change From Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Performance Subscale
Description: The TETRAS is an essential tremor and activities of daily living rating scale. The full scale has 2 sections, the Performance subscale (PS) and the ADL subscale. The PS consists of 9 items covering different body regions. These 9 items are rated on a 5-point scale (ranging from 0 to 4). One item, Item 4, consists of ratings for 3 tasks rated separately for upper limbs on both sides of the body for a total of 6 ratings. The total score of the 9 items (14 ratings) ranges from 0 to 70 with higher scores indicating greater tremor severity. The total score and individual item ratings will be evaluated as outcomes in this trial. Baseline is defined as the last non-missing value collected prior to receiving first dose of study drug.
Time Frame: Baseline (Day 0), Days 7 and 14
Population: FAS population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part A: PRAX-944 20mg to 40mg OLT
Number analyzed (Participants) | 6
scores on a scale
  Change from baseline to Day 7 | -1.990 [-7.5467 to 3.5672]
  Change from baseline to Day 14 | -5.163 [-11.1371 to 0.8108]
Statistical Analysis 1: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.4025, Mixed Models Analysis; Change from baseline to Day 7
Statistical Analysis 2: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.0766, Mixed Models Analysis — Change from baseline to Day 14

6. Secondary Outcome: Part A: Change From Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Upper Limb Score Measured by Accelerometry
Description: Accelerometer was used to evaluate record coordinates and accelerations in the 3D space over time. The 3 maneuvers in the upper limb item will be completed for both arms, first for the right arm and then for the left. Each upper limb sub-item is scored on a scale from 0 to 4 including to 0.1 increments. The accelerometer upper limb total score, ranges from 0 to 24. A decrease in score is indicative of improvement. Baseline is defined as the last non-missing value collected prior to receiving first dose of study drug. Change from baseline will be defined as assessment value minus baseline value.
Time Frame: Baseline (Day 0), Days 7 and 14
Population: FAS Population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part A: PRAX-944 20mg to 40mg OLT
Number analyzed (Participants) | 3
scores on a scale
  Change from baseline to Day 7 | -1.100 [-3.3733 to 1.1733]
  Change from baseline to Day 14 | -1.300 [-3.5733 to 0.9733]
Statistical Analysis 1: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.2501, Mixed Models Analysis — Change from baseline to Day 7
Statistical Analysis 2: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.1874, Mixed Models Analysis — Chnage from baseline to Day 14

7. Secondary Outcome: Part A: Change From Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Performance Subscale Individual Items # 6 (Spiral Drawing) and Items #7 (Handwriting)
Description: The TETRAS ADL subscale is a 12-item assessment of typical daily activities that are impacted by tremor. Activities are assessed in the following functional domains: speaking, feeding, drinking, personal hygiene, dressing, writing, and social activity. The impact to each function is rated on a 5-point Likert scale from 0 to 4. The ADL subscale score is calculated as the sum of all 12 items and ranges from 0 to 48 with higher scores reflecting higher impact. Baseline is defined as the last non-missing value collected prior to receiving first dose of study drug. Change from baseline will be defined as assessment value minus baseline value.
Time Frame: Baseline (Day 0), Days 7 and 14
Population: FAS population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part A: PRAX-944 20mg to 40mg OLT
Number analyzed (Participants) | 6
scores on a scale
  Item 6 Archimedes Spiral (Right) Change from baseline to Day 7 | -0.091 [-0.5713 to 0.389]
  Item 6 Archimedes Spiral (Left) Change from baseline to Day 7 | -0.213 [-1.2762 to 0.8501]
  Item 7 Handwriting Change from baseline to Day 7 | -0.012 [-0.7215 to 0.6975]
  Item 7 Handwriting Change from baseline to Day 14 | -0.348 [-1.0966 to 0.4013]
  Item 6 Archimedes Spiral (Right) Change from baseline to Day 14 | -0.346 [-0.9765 to 0.2836]
  Item 6 Archimedes Spiral (Left) Change from baseline to Day 14 | -0.468 [-1.3845 to 0.4487]
Statistical Analysis 1: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.4722, Mixed Models Analysis — Item 6 Archimedes Spiral (right) change from baseline to Day 7
Statistical Analysis 2: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.6215, Mixed Models Analysis — Item 6 Archimedes Spiral (left) change from baseline to Day 7
Statistical Analysis 3: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.9648, Mixed Models Analysis — Item 7 Handwriting change from baseline to Day 7
Statistical Analysis 4: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.2855, Mixed Models Analysis — Item 7 Handwriting change from baseline to Day 14
Statistical Analysis 5: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.2050, Mixed Models Analysis — Item 6 Archimedes Spiral (right) change from baseline to Day 14
Statistical Analysis 6: Comparison: Part A: PRAX-944 20mg to 40mg OLT; Test type: Other; p = 0.2364, Mixed Models Analysis — Item 6 Archimedes Spiral (left) change from baseline to Day 14

8. Secondary Outcome: Part A: Number of Participants With Adverse Events (AE), Related AE, and AE Leading to Treatment Discontinuation
Description: as for outcome 2
Time Frame: Up to Day 21
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Part A: PRAX-944 20mg to 40mg OLT
Number analyzed (Participants) | 7
participants
  Any AE | 6
  Related AE | 4
  AE Leading to Treatment Discontinuation | 1
  Mild AE | 6
  Moderate AE | 1
  Severe AE | 0

9. Secondary Outcome: Part A: Number of Participants With Clinically Significant Abnormalities in Vital Signs, Laboratory Values and Electrocardiogram Parameters
Description: as for outcome 3
Time Frame: Up to Day 21
Population: Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Part A: PRAX-944 20mg to 40mg OLT
Number analyzed (Participants) | 7
Participants | 0

10. Secondary Outcome: Part A: Number of Participants With Suicidal Ideation or Behavior Assessed Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: as for outcome 4
Time Frame: Up to Day 21
Population: Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Part A: PRAX-944 20mg to 40mg OLT
Number analyzed (Participants) | 7
Participants | 0

11. Secondary Outcome: Part B: Change From Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Upper Limb Score During OLT Phase
Description: as for outcome 1
Time Frame: Baseline (Day 0) and Day 42
Population: FAS Population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT
Number analyzed (Participants) | 11
scores on a scale | -2.090 [-3.8223 to -0.3585]
Statistical Analysis 1: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0216, Mixed Models Analysis

12. Secondary Outcome: Part B: Change From Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Upper Limb Score During OLT Phase
Description: as for outcome 1
Time Frame: Baseline (Day 0), Days 7 and 21
Population: FAS. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT
Number analyzed (Participants) | 12
scores on a scale
  Change from baseline to Day 7: number analyzed (Participants) | 10
  Change from baseline to Day 7 | -0.967 [-2.1795 to 0.2447]
  Change from baseline to Day 21 | -1.143 [-2.1269 to -0.1598]
Statistical Analysis 1: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.1042, Mixed Models Analysis — Change from baseline Day 7
Statistical Analysis 2: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0257, Mixed Models Analysis — Change from baseline Day 21

13. Secondary Outcome: Part B: Change From Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Performance Subscale During OLT Phase
Description: TETRAS Performance Subscale was used to assess essential tremor as scored by the independent video raters. The performance subscale consists of 9 items, i.e. item 1 (head), item 2 (face), item 3 (voice), each of the 6 sub-items for item 4 (upper limb), the maximum of the 4 sub-items for item 5 (lower limb), 2 sub-items (right and left side) for item 6 (Archimedes spirals), item 7 (handwriting), 2 sub-items (right and left side) for item 8 (dot approximation), and item 9 (standing) for a total score ranging from 0 to 64 from 16 sub-items. Each item is rated on a scale of 0 to 4, including 0.5 increments. A lower score is indicative of improvement. The total score has been presented. Baseline is defined as the last non-missing value collected prior to receiving first dose of study drug. Change from baseline will be defined as assessment value minus baseline value.
Time Frame: Baseline (Day 0) and Days 7, 21 and 42
Population: FAS population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT
Number analyzed (Participants) | 12
scores on a scale
  Change from baseline to Day 7: number analyzed (Participants) | 10
  Change from baseline to Day 7 | -1.253 [-3.8185 to 1.3133]
  Change from baseline to Day 21 | -1.449 [-3.7708 to 0.8734]
  Change from baseline to Day 42: number analyzed (Participants) | 11
  Change from baseline to Day 42 | -2.771 [-6.2554 to 0.7127]
Statistical Analysis 1: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.2971, Mixed Models Analysis — Change from baseline to Day 7
Statistical Analysis 2: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.2034, Mixed Models Analysis — Change from baseline Day 21
Statistical Analysis 3: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.1105, Mixed Models Analysis — Change from baseline to Day 42

14. Secondary Outcome: Part B: Change From Baseline in Essential Tremor Rating Assessment Scale (TETRAS) Upper Limb Score Measured by Accelerometry During OLT Phase
Description: as for outcome 6
Time Frame: Baseline (Day 0), and Days 7, 21 and 42
Population: FAS population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT
Number analyzed (Participants) | 11
scores on a scale
  Change from baseline to Day 7: number analyzed (Participants) | 10
  Change from baseline to Day 7 | -1.235 [-2.0318 to -0.4376]
  Change from baseline to Day 21 | -1.835 [-2.8523 to -0.8179]
  Change from baseline to Day 42 | -1.766 [-2.9106 to -0.6223]
Statistical Analysis 1: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0050, Mixed Models Analysis — Change from baseline to Day 7
Statistical Analysis 2: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0018, Mixed Models Analysis — Change from baseline to Day 21
Statistical Analysis 3: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0061, Mixed Models Analysis — Change from baseline to Day 42

15. Secondary Outcome: Part B: Change From Baseline in TETRAS Performance Subscale Individual Items # 6 (Spiral Drawing) and Items #7 (Handwriting)
Description: TETRAS Performance Subscale was used to assess essential tremor as scored by the independent video raters. The performance subscale consists of 9 items, i.e. item 1 (head), item 2 (face), item 3 (voice), each of the 6 sub-items for item 4 (upper limb), the maximum of the 4 sub-items for item 5 (lower limb), 2 sub-items (right and left side) for item 6 (Archimedes spirals), item 7 (handwriting), 2 sub-items (right and left side) for item 8 (dot approximation), and item 9 (standing) for a total score ranging from 0 to 64 from 16 sub-items. Each item is rated on a scale of 0 to 4, including 0.5 increments. A lower score is indicative of improvement. Baseline is defined as the last non-missing value collected prior to receiving first dose of study drug. Change from baseline will be defined as assessment value minus baseline value.
Time Frame: Baseline (Day 0), Days 7, 21 and 42
Population: FAS Population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT
Number analyzed (Participants) | 12
scores on a scale
  Item#6 Archimedes spirals (right) Change from baseline to Day 7: number analyzed (Participants) | 10
  Item#6 Archimedes spirals (right) Change from baseline to Day 7 | 0.006 [-0.4387 to 0.4500]
  Item#6 Archimedes spirals (left) Change from baseline to Day 7 | 0.221 [-0.1329 to 0.5739]
  Item#7 Handwriting Change from baseline to Day 7 | -0.019 [-0.6477 to 0.6087]
  Item#6 Archimedes spirals (right) Change from baseline to Day 21 | -0.240 [-0.5006 to 0.0202]
  Item#6 Archimedes spirals (left) Change from baseline to Day 21 | -0.012 [-0.2547 to 0.2316]
  Item#7 Handwriting Change from baseline to Day 21 | 0.107 [-0.3613 to 0.5745]
  Item#6 Archimedes spirals (right) Change from baseline to Day 42 | -0.239 [-0.6711 to 0.1930]
  Item#6 Archimedes spirals (left) Change from baseline to Day 42 | -0.072 [-0.4488 to 0.3044]
  Item#7 Handwriting Change from baseline to Day 42 | -0.054 [-0.6984 to 0.5911]
Statistical Analysis 1: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.9776, Mixed Models Analysis — Item 6 Archimedes Spiral (right) change from baseline to Day 7
Statistical Analysis 2: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.1962, Mixed Models Analysis — Item 6 Archimedes Spiral (left) change from baseline to Day 7
Statistical Analysis 3: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.9419, Mixed Models Analysis — Item 7 Handwriting change from baseline to Day 7
Statistical Analysis 4: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0668, Mixed Models Analysis — Item 6 Archimedes Spiral (right) change from baseline to Day 21
Statistical Analysis 5: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.9191, Mixed Models Analysis — Item 6 Archimedes Spiral (left) change from baseline to Day 21
Statistical Analysis 6: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.6075, Mixed Models Analysis — Item 7 Handwriting change from baseline to Day 21
Statistical Analysis 7: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.2460, Mixed Models Analysis — Item 6 Archimedes Spiral (right) change from baseline to Day 42
Statistical Analysis 8: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.6736, Mixed Models Analysis — Item 6 Archimedes Spiral (left) change from baseline to Day 42
Statistical Analysis 9: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.8511, Mixed Models Analysis — Item 7 Handwriting change from baseline to Day 42

16. Secondary Outcome: Part B: Change From Baseline in TETRAS Activities of Daily Living (ADL) Score
Description: as for outcome 7
Time Frame: Baseline (Day 0), Days 7, 21 and 42
Population: FAS population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT
Number analyzed (Participants) | 12
scores on a scale
  Change from baseline to Day 7: number analyzed (Participants) | 10
  Change from baseline to Day 7 | -1.986 [-4.8142 to 0.8417]
  Change from baseline to Day 21 | -3.475 [-7.0260 to 0.0756]
  Change from baseline to Day 42: number analyzed (Participants) | 11
  Change from baseline to Day 42 | -8.207 [-12.5655 to -3.8481]
Statistical Analysis 1: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.1505, Mixed Models Analysis — Change from baseline to Day 7
Statistical Analysis 2: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0543, Mixed Models Analysis — Change from baseline to Day 21
Statistical Analysis 3: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0015, Mixed Models Analysis — Change from baseline to Day 42

17. Secondary Outcome: Part B: Change From Baseline in Quality of Life in Essential Tremor Questionnaire (QUEST) Total Scores.
Description: Quality of Life in Essential Tremor Questionnaire (QUEST) is a patient-reported ET-specific 30-item, specific quality of life scale. Items contribute to five dimensions. Physical/ADL (9 items ), Psychosocial (9 items), Communication (3 items), Hobbies/Leisure (3 items), and Work/Finances (6 items). The QUEST total and subscale scores are calculated as the sum of all applicable items divided by the number of applicable items times 100. Higher score indicates greater dissatisfaction with that domain of QOL. Maximal score 100: worse quality of life. Minimal Score 0: best quality of life. Baseline is defined as the last non-missing value collected prior to receiving first dose of study drug. Change from baseline will be defined as assessment value minus baseline value.
Time Frame: Baseline (Day 0), Days 7, 21 and 42
Population: FAS population. Only those participants with data available at indicated timepoints have been presented.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Part B: PRAX-944 20mg to 120mg OLT
Number analyzed (Participants) | 10
scores on a scale
  Change from baseline to Day 7: number analyzed (Participants) | 8
  Change from baseline to Day 7 | -0.561 [-7.7823 to 6.6611]
  Change from baseline to Day 21 | -5.933 [-12.1961 to 0.3310]
  Change from baseline to Day 42: number analyzed (Participants) | 9
  Change from baseline to Day 42 | -8.203 [-17.9048 to 1.4991]
Statistical Analysis 1: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.8638, Mixed Models Analysis — Change from baseline to Day 7
Statistical Analysis 2: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0605, Mixed Models Analysis — Change from baseline to Day 21
Statistical Analysis 3: Comparison: Part B: PRAX-944 20mg to 120mg OLT; Test type: Other; p = 0.0871, Mixed Models Analysis — Change from baseline to Day 42

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to Day 70 (up to Day 21 for Part A and up to Day 70 for Part B)
Description: All Adverse Events were collected from the time the participant provided consent to participate in the study until the end of the study (last study visit) for the participant.
Arm/Group | Part A: PRAX-944 20mg to 40mg Open-Label Titration (OLT) | Part B: PRAX-944 20mg to 120mg OLT | Part B: PRAX-944 120mg Randomized Withdrawal Phase (RWD) | Part B: Placebo RWD
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/17 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/17 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 6/7 | 15/17 | 1/6 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: PRAX-944 20mg to 40mg Open-Label Titration (OLT) (N=7) | Part B: PRAX-944 20mg to 120mg OLT (N=17) | Part B: PRAX-944 120mg Randomized Withdrawal Phase (RWD) (N=6) | Part B: Placebo RWD (N=5)
Cyst (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: PRAX-944 20mg to 40mg Open-Label Titration (OLT) (N=7) | Part B: PRAX-944 20mg to 120mg OLT (N=17) | Part B: PRAX-944 120mg Randomized Withdrawal Phase (RWD) (N=6) | Part B: Placebo RWD (N=5)
Photophobia (Eye disorders) | 0 | 1 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 (0) | 6 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Cyst (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 4 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 6 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0
Essential tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucinations, mixed (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0 | 0
Initial Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Middle Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to repeated mistakes during the eligibility review process, a Corrective and Preventative Actions (CAPA) report was issued and enrollment at one site was suspended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT05021978/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT05021978/SAP_001.pdf